CLINICAL TRIAL: NCT05670561
Title: Effects of Esketamine on Acute Abdominal Pain After TACE in Patients With Hepatocellular Carcinoma:a Prospective Study TACE(Transcatheter Arterial Chemoembolization)
Brief Title: Effects of Esketamine on Acute Abdominal Pain After TACE in Patients With Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: pain after TACE
Record Dates: First submitted 2023-01-02; First posted 2023-01-04 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-02

CONDITIONS: Hepatocellular Carcinoma; Transcatheter Arterial Chemoembolization; Pain
MeSH Terms: conditions — Carcinoma, Hepatocellular; Pain | interventions — Esketamine; Sufentanil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Esketamine-PCIA(patient controlled intravenous analgesia) (Experimental): PCIA formula#100ml analgesic solution was prepared by adding 2.5 mg/kg Esketamine and 8mg ondansetron into normal saline.
  Interventions: Drug: Esketamine
- Sufentanil-PCIA(patient controlled intravenous analgesia) (Active Comparator): PCIA formula#100ml analgesic solution was prepared by adding 2 μ g/kg sufentanil and 8mg ondansetron into normal saline.
  Interventions: Drug: Sufentanil

INTERVENTIONS:
Drug: Esketamine — PCIA formula#100ml analgesic solution was prepared by adding 2.5 mg/kg Esketamine and 8mg ondansetron into normal saline. 30min before TACE treatment, the first dose of 2ml was slowly injected intravenously. No obvious adverse reactions were observed for 10min.The PCIA pump was commenced at the beginning of TACE. Parameter setting of intravenous analgesia pump: the total volume is 100ml; The duration is 2ml / h; The single dose is 2ml each time; The limit quantity is 10ml / h; The locking time was 10min and the analgesia lasted for 48h. The target value of analgesia in this study was NRS (Numerical Rating Scale)< 4; If NRS ≥ 4, when the effect is still poor after adding drugs by pressing the analgesic pump, the investigators will give the remedial drug(dolantin 50mg im st) according to the patient's condition.
  Other Names: patient controlled intravenous analgesia
  Arms: Esketamine-PCIA(patient controlled intravenous analgesia)
Drug: Sufentanil — PCIA formula#100ml analgesic solution was prepared by adding 2 μ g/kg sufentanil and 8mg ondansetron into normal saline. 30min before TACE treatment, the first dose of 2ml was slowly injected intravenously.No obvious adverse reactions were observed for 10min. The PCIA pump was commenced at the beginning of TACE. Parameter setting of intravenous analgesia pump: the total volume is 100ml; The duration is 2ml / h; The single dose is 2ml each time; The limit quantity is 10ml / h; The locking time was 10min and the analgesia lasted for 48h. The target value of analgesia in this study was NRS (Numerical Rating Scale)< 4; If NRS ≥ 4, when the effect is still poor after adding drugs by pressing the analgesic pump, the investigators will give the remedial drug(dolantin 50mg im st) according to the patient's condition.
  Other Names: patient controlled intravenous analgesia
  Arms: Sufentanil-PCIA(patient controlled intravenous analgesia)

SUMMARY:
Pain is the main complication after TACE(Transcatheter Arterial Chemoembolization) for hepatocellular carcinoma, and its pathogenesis is not clear.The pain may be related to partial liver tissue swelling after blocking the tumor blood supply artery embolization agent, transient hepatic swelling causing tension or strain on the liver capsule, and chemical irritation by the anticancer drug-Lipiodol mixture,the inadvertent embolization of normal organs and individual sensitivity to pain. Ketamine produces anesthetic and analgesic effects mainly by inhibiting NMDA receptor(N-methyl-D-aspartic acid receptor), and previous studies have shown that low concentrations of ketamine have obvious analgesic effects. Not only that, ketamine also produces analgesic effects by inhibiting opioid receptors via G-protein coupling. In addition, ketamine can bind to monoaminergic receptors in the central and peripheral nervous system, showing an anticholinergic effect and producing an antispasmodic effect. Ketamine also inhibits inflammatory pain by reducing nitric oxide production by inhibiting nitric oxide synthase. Esketamine is about three to four times more potent than ketamine. Therefore,esketamine requires a lower dose, about half the dose of ketamine, to produce anesthetic and analgesic effects, with fewer side effects.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 80
* Participate in this study and sign informed consent
* Voluntarily receive preoperative intravenous analgesia
* Patients receiving TACE treatment
* HCC (hepatocellular carcinoma)patients with primary liver cancer BCLC(Barcelona Clinic Liver Cancer) stage A-C, liver function A-B

Exclusion Criteria:

* Patients who were unable to cooperate or refused to participate in the trial
* Pregnant women
* Patients with or having a history of serious mental disorders
* Patients with poorly controlled or untreated hypertension (arterial hypertension, resting systolic / diastolic blood pressure more than 180/100mg)
* Patients with unstable angina pectoris or myocardial infarction within 6 months or congestive heart failure
* Patients with intracranial hypertension or glaucoma
* Patients with hyperthyroidism without treatment or insufficient treatment
* Patients with severe respiratory dysfunction
* Allergy or existing contraindication to chemotherapeutic drugs, opioids or ketamine drugs

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-05 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity at 4hours after the beginning of TACE operation | From 0 to 4hours after the beginning of TACE
  Pain intensity is assessed by numerical rating scale pain scores(0-10,0 represents painless,10 represents intolerable pain;higher scores mean a worse outcome)
Pain Intensity at 8hours after the beginning of TACE operation | From 4hours to 8hours after the beginning of TACE operation
  Pain intensity is assessed by numerical rating scale pain scores(0-10,0 represents painless,10 represents intolerable pain;higher scores mean a worse outcome)
Pain Intensity at 12hours after the beginning of TACE operation | From 8hours to 12hours after the beginning of TACE operation
  Pain intensity is assessed by numerical rating scale pain scores(0-10,0 represents painless,10 represents intolerable pain;higher scores mean a worse outcome)

SECONDARY OUTCOMES:
Pain Intensity at 18hours after the beginning of TACE operation | From 12hours to 18hours after the beginning of TACE operation
  Pain intensity is assessed by numerical rating scale pain scores(0-10,0 represents painless,10 represents intolerable pain;higher scores mean a worse outcome)
Pain Intensity at 24hours after the beginning of TACE operation | From 18hours to 24hours after the beginning of TACE operation
  Pain intensity is assessed by numerical rating scale pain scores(0-10,0 represents painless,10 represents intolerable pain;higher scores mean a worse outcome)
Pain Intensity at 30hours after the beginning of TACE operation | From 24hours to 30hours after the beginning of TACE operation
  Pain intensity is assessed by numerical rating scale pain scores(0-10,0 represents painless,10 represents intolerable pain;higher scores mean a worse outcome)
Pain Intensity at 36hours after the beginning of TACE operation | From 30hours to 36hours after the beginning of TACE operation
  Pain intensity is assessed by numerical rating scale pain scores(0-10,0 represents painless,10 represents intolerable pain;higher scores mean a worse outcome)
Pain Intensity at 42hours after the beginning of TACE operation | From 36hours to 42hours after the beginning of TACE operation
  Pain intensity is assessed by numerical rating scale pain scores(0-10,0 represents painless,10 represents intolerable pain;higher scores mean a worse outcome)
Pain Intensity at 48hours after the beginning of TACE operation | From 42hours to 48hours after the beginning of TACE operation
  Pain intensity is assessed by numerical rating scale pain scores(0-10,0 represents painless,10 represents intolerable pain;higher scores mean a worse outcome)
Maximum Pain Intensity in the First 4hours after the beginning of TACE operation | From the beginning of TACE operation to 4hours after the beginning of TACE operation
  Pain intensity is assessed by numerical rating scale pain scores(0-10,0 represents painless,10 represents intolerable pain;higher scores mean a worse outcome)
Maximum Pain Intensity in the Second 4hours after the beginning of TACE operation | From 4hours to 8hours after the beginning of TACE operation
  Pain intensity is assessed by numerical rating scale pain scores(0-10,0 represents painless,10 represents intolerable pain;higher scores mean a worse outcome)
Maximum Pain Intensity in the Third 4hours after the beginning of TACE operation | From 8hours to 12hours after the beginning of TACE operation
  Pain intensity is assessed by numerical rating scale pain scores(0-10,0 represents painless,10 represents intolerable pain;higher scores mean a worse outcome)
Analgesic Consumption | From 0 to 48 hours after the beginning of TACE operation
  Analgesic consumption is assessed by the total amount of pain remedy with dolantin when the analgesic effect is poor.

OTHER OUTCOMES:
Ramsay Sedation Score at 1 hour after the beginning of TACE operation | From 0 to 1hour after the beginning of TACE operation
  Grade 1 (soberness- the patient is anxious, uneasy or irritable)# Grade 2 (soberness- the patient is cooperative, has good orientation or is quiet)# Grade 3 (soberness- the patient only responds to commands)# Grade 4 (sleep-the patient responds quickly to light tapping between eyebrows or strong sound stimulation)# Grade 5 (sleep-the patient responds slowly to light tapping between the eyebrows or strong sound stimulation) and Grade 6 (sleep-the patient has no response to light tapping between eyebrows or strong sound stimulation). Grade 1 indicates no sedation ; Grade 2 and 3 indicate good sedation ; Grade 4 to 6 indicate poor sedation.
Ramsay Sedation Score at 2 hours after the beginning of TACE operation | From 1hour to 2hours after the beginning of TACE operation
  Grade 1 (soberness- the patient is anxious, uneasy or irritable)# Grade 2 (soberness- the patient is cooperative, has good orientation or is quiet)# Grade 3 (soberness- the patient only responds to commands)# Grade 4 (sleep-the patient responds quickly to light tapping between eyebrows or strong sound stimulation)# Grade 5 (sleep-the patient responds slowly to light tapping between the eyebrows or strong sound stimulation) and Grade 6 (sleep-the patient has no response to light tapping between eyebrows or strong sound stimulation). Grade 1 indicates no sedation ; Grade 2 and 3 indicate good sedation ; Grade 4 to 6 indicate poor sedation.
Ramsay Sedation Score at 3 hours after the beginning of TACE operation | From 2hours to 3hours after the beginning of TACE operation
  Grade 1 (soberness- the patient is anxious, uneasy or irritable)# Grade 2 (soberness- the patient is cooperative, has good orientation or is quiet)# Grade 3 (soberness- the patient only responds to commands)# Grade 4 (sleep-the patient responds quickly to light tapping between eyebrows or strong sound stimulation)# Grade 5 (sleep-the patient responds slowly to light tapping between the eyebrows or strong sound stimulation) and Grade 6 (sleep-the patient has no response to light tapping between eyebrows or strong sound stimulation). Grade 1 indicates no sedation ; Grade 2 and 3 indicate good sedation ; Grade 4 to 6 indicate poor sedation.
The Quality of Sleep on the Day Just before TACE Treatment | From the day just before TACE treatment to the operation day
  The Richards-Campbell Sleep Questionnaire (RCSQ) is assessed by the quality of patients' sleep quality.0~25 points indicate poor sleep quality;76~100 points indicate good sleep quality (0-100, 0 represents the worst sleep quality; 100 represents the best sleep quality ;higher scores mean a better outcome)
The Quality of Sleep on the Operation Day | From the operation day to first day after TACE treatment
  The Richards-Campbell Sleep Questionnaire (RCSQ) is assessed by the quality of patients' sleep quality.0~25 points indicate poor sleep quality;76~100 points indicate good sleep quality (0-100, 0 represents the worst sleep quality; 100 represents the best sleep quality ;higher scores mean a better outcome)
The Quality of Sleep on the First Day after TACE Treatment | From the first day after TACE treatment to the second day after TACE treatment
  The Richards-Campbell Sleep Questionnaire (RCSQ) is assessed by the quality of patients' sleep quality.0~25 points indicate poor sleep quality;76~100 points indicate good sleep quality (0-100, 0 represents the worst sleep quality; 100 represents the best sleep quality ;higher scores mean a better outcome)
Adverse Reaction | From 0 to 48 hours after the beginning of TACE operation
  Adverse reaction is recorded according to follow-up visits after TACE treatment
Degree of Satisfaction | From 0 to 24 hours after the beginning of TACE operation
  Degree of satisfaction is assessed by patient using numerical rating scale (0-10, 0 represents unsatisfactory; 10 represents complete satisfaction;higher scores mean a better outcome)
Quality-of-Life Assessment at the the beginning of TACE operation | From the beginning of TACE operation to 0 hour after the beginning of TACE operation
  Quality-of-life contains patients' quality of sleep，fatigue, spiritual well-being, and appetite.The scores were categorized as follows: 1，worst；2，bad；3， mild；4， normal；5，very good.
Quality-of-Life Assessment at 24hours after the beginning of TACE operation | From 0 to 24 hours after the beginning of TACE operation
  Quality-of-life contains patients' quality of sleep，fatigue, spiritual well-being, and appetite.The scores were categorized as follows: 1，worst；2，bad；3， mild；4， normal；5，very good.

CONTACTS AND LOCATIONS:
Overall Officials: Huang He, MD, Study Chair — The Second Affiliated Hospital, Chongqing Medical University
Locations (1):
- The Second Affiliated Hospital, Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data for this study is available from the sponsor on reasonable request through email.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: Within one year